CLINICAL TRIAL: NCT00700765
Title: Observational, Safety Study in Subjects Using Levemir® (Insulin Detemir) for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes Mellitus
Brief Title: Observational Study to Evaluate Safety of Levemir® in Type 1 and Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3528
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — For study drug, start dose and frequency of administration to be prescribed by the physician as a result of normal clinical evaluation
  Other Names: Levemir®

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the incidence of adverse events while using Levemir® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus

Exclusion Criteria:

* Subjects who are unlikely to comply with the protocol
* Subjects who are currently being treated with Levemir®
* Subjects who previously were enrolled into the study
* Subjects with hypersensitivity to Levemir® or any of its excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 1 or type 2 diabetes who is prescribed insulin detemir at the physician's discretion
Sampling Method: Non-Probability Sample
Enrollment: 1531 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions (SADRs) | during treatment
Major hypoglycaemic events | during treatment

SECONDARY OUTCOMES:
Number of serious adverse events | during treatment
Number of all adverse events | during treatment
Number of all hypoglycaemic events | the last 4 weeks of treatment
Weight changes | after 12 weeks
HbA1c | after 12 weeks and 26 weeks of treatment
Variability in fasting blood glucose (FBG) and average plasma glucose level | after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com